CLINICAL TRIAL: NCT02935413
Title: Combined tDCS and Vision Restoration Training in Subacute Stroke Rehabilitation: A Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: Neurologisches Therapiezentrum Gmundnerberg (Other)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Professor, University of Magdeburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CES_NTG_Pilot
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Hemianopia; Stroke
MeSH Terms: conditions — Hemianopsia; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS (Active Comparator): group receiving complete treatment of transcranial direct current stimulation
  Interventions: Device: tDCS
- Standard rehabilitation (Active Comparator): Standard rehabilitation procedures
  Interventions: Behavioral: Standard rehabilitation

INTERVENTIONS:
Device: tDCS — Device: verum tDCS real transcranial direct current stimulation,10 sessions, 2mA for 20 minutes Behavioral: VRT Vision restoration training, 10 sessions, 20 minutes
  Arms: tDCS
Behavioral: Standard rehabilitation — Standard rehabilitation procedures involving PC-based training of saccades and visual exploration
  Arms: Standard rehabilitation

SUMMARY:
The purpose of this Study is to determine whether non-invasive transcranial direct current stimulation (tDCS) is effective in increasing rehabilitation effects after stroke in visual Cortex.

DETAILED DESCRIPTION:
Visual field defects after posterior cerebral artery stroke can be improved by vision restoration training (VRT), but when combined with transcranial direct current stimulation (tDCS) which alters brain excitability, vision restoration can be potentiated in the chronic stage. Because it is possible that such therapy may be more effective during the early recovery phase after the stroke and can reach patients during the rehabilitation phase, investigators wished to explore the applicability, efficacy and safety of early intervention with a combined tDCS/VRT treatment.

Seven post-acute stroke homonymous hemianopia patients were assigned to 10 sessions of combined tDCS (2mA, 10 daily sessions of 15-20 min) and VRT. The primary outcome criterion was the pre-post change in perimetric detection thresholds in percent. The results were compared to 7 age and stroke lesion matched controls of our patient data pool who received standard rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Posterior Cerebral Artery Stroke
* Visual Field Defect
* Lesion age 4 weeks up to 6 month max

Exclusion Criteria:

* Electrical Implants
* Metal artefacts in head
* Epilepsy
* Visual Neglect

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change of mean sensitivity (in dB) detection threshold from baseline to post-intervention | 14-20 days post treatment,

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Alber, MS, Principal Investigator — Neurologisches Therapiezentrum Gmundnerberg
Locations (2):
- Neurologisches Therapiezentrum Gmundnerberg, Altmünster, Austria
- Inst. f. Medical Psychology, Univ. of Magdeburg, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alber R, Moser H, Gall C, Sabel BA. Combined Transcranial Direct Current Stimulation and Vision Restoration Training in Subacute Stroke Rehabilitation: A Pilot Study. PM R. 2017 Aug;9(8):787-794. doi: 10.1016/j.pmrj.2016.12.003. Epub 2017 Jan 8. PMID 28082176